CLINICAL TRIAL: NCT06603571
Title: A Phase 2, Parallel-Group, Double-Blind, Placebo-Controlled Study to Investigate Weight Management With LY3841136 and Tirzepatide, Alone or in Combination, in Adult Participants With Obesity or Overweight With Type 2 Diabetes
Brief Title: A Study to Investigate Weight Management With LY3841136 and Tirzepatide (LY3298176), Alone or in Combination, in Adult Participants With Obesity or Overweight With Type 2 Diabetes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18809; W8M-MC-LAA2 (Other: Eli Lilly and Company); W8M-MC-CWMM Master Protocol (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Overweight
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- LY3841136 Dose 1 (Experimental): Participants will receive LY3841136 subcutaneously (SC)
  Interventions: Drug: LY3841136
- LY3841136 Dose 2 (Experimental): Participants will receive LY3841136 SC
  Interventions: Drug: LY3841136
- LY3841136 Dose 3 (Experimental): Participants will receive LY3841136 SC
  Interventions: Drug: LY3841136
- LY3841136 Dose 1 + Tirzepatide Dose 1 (Experimental): Participants will receive LY3841136 SC and Tirzepatide SC
  Interventions: Drug: LY3841136; Drug: Tirzepatide
- LY3841136 Dose 2 + Tirzepatide Dose 1 (Experimental): Participants will receive LY3841136 SC and Tirzepatide SC
  Interventions: Drug: LY3841136; Drug: Tirzepatide
- LY3841136 Dose 2 + Tirzepatide Dose 2 (Experimental): Participants will receive LY3841136 SC and Tirzepatide SC
  Interventions: Drug: LY3841136; Drug: Tirzepatide
- LY3841136 Dose 3 + Tirzepatide Dose 3 (Experimental): Participants will receive LY3841136 SC and Tirzepatide SC
  Interventions: Drug: LY3841136; Drug: Tirzepatide
- Tirzepatide Dose 3 (Active Comparator): Participants will receive Tirzepatide SC
  Interventions: Drug: Tirzepatide
- LY3841136 Dose 2 + Tirzepatide Dose 3 (Experimental): Participants will receive LY3841136 SC and Tirzepatide SC
  Interventions: Drug: LY3841136; Drug: Tirzepatide
- Placebo (Placebo Comparator): Participants will receive placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3841136 — Administered SC
  Arms: LY3841136 Dose 1; LY3841136 Dose 1 + Tirzepatide Dose 1; LY3841136 Dose 2; LY3841136 Dose 2 + Tirzepatide Dose 1; LY3841136 Dose 2 + Tirzepatide Dose 2; LY3841136 Dose 2 + Tirzepatide Dose 3; LY3841136 Dose 3; LY3841136 Dose 3 + Tirzepatide Dose 3
Drug: Tirzepatide — Administered SC
  Arms: LY3841136 Dose 1 + Tirzepatide Dose 1; LY3841136 Dose 2 + Tirzepatide Dose 1; LY3841136 Dose 2 + Tirzepatide Dose 2; LY3841136 Dose 2 + Tirzepatide Dose 3; LY3841136 Dose 3 + Tirzepatide Dose 3; Tirzepatide Dose 3
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study, performed under the master protocol W8M-MC-CWMM (NCT06143956), is to investigate the safety and efficacy of LY3841136 for chronic weight management alone or in combination with Tirzepatide across a wide dose range in participants with Type 2 Diabetes. Participation in the study will last about 64 weeks.

ELIGIBILITY:
Inclusion Criteria:

W8M-MC-LAA2

* Have a Body Mass Index (BMI) of ≥27 kilograms per square meter (kg/m²)
* Have Type 2 Diabetes
* Have a HbA1c ≥7.0 % (53 millimoles/mole (mmol/mol)) to ≤10.5% (91 mmol/mol) and treated with diet and exercise alone or with a stable dose of metformin (and not more than the locally approved dose) with or without a sodium-glucose cotransporter 2 (SGLT2) inhibitor for at least 3 months prior to screening

W8M-MC-CWMM:

* Have had a stable body weight for the 3 months prior to randomization (<5% body weight gain and/or loss)

Exclusion Criteria:

W8M-MC-LAA2

* Have a history of severe hypoglycemia or hypoglycemia unawareness within the last 6 months prior to screening
* Have an on-going or history of bradyarrhythmia and/or sinus bradycardia
* Have an elevated resting pulse rate (mean >100 beats per minute (bpm)) or reduced resting pulse rate (mean <60 bpm) at screening
* Have any of the following cardiovascular conditions within 6 months prior to screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * unstable angina, or
  * hospitalization due to congestive heart failure
* Have renal impairment measured as estimated glomerular filtration rate (eGFR) <45 milliliters per minute (mL/min)/1.73 m2
* Have a history of acute or chronic pancreatitis
* Have fasting triglycerides >500 milligrams per deciliter (mg/dL) (5.7 mmol/L) at screening
* All concomitant medications should be at a stable dose for at least 3 months prior to screening

W8M-MC-CWMM

* Have a prior or planned surgical treatment for obesity, except prior liposuction or abdominoplasty, if performed >1 year prior to screening.
* Have type 1 diabetes mellitus, latent autoimmune diabetes in adults, or history of ketoacidosis or hyperosmolar coma.
* Have poorly controlled hypertension.
* Have a history of symptomatic gallbladder disease within the past 2 years
* Have signs and symptoms of any liver disease other than nonalcoholic fatty liver disease.
* Have a lifetime history of suicide attempts.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 48

SECONDARY OUTCOMES:
Change from Baseline in Body Weight | Baseline, Week 48
Percentage of Participants Who Achieve ≥5% Body Weight Reduction | Week 48
Percentage of Participants Who Achieve ≥10% Body Weight Reduction | Week 48
Change from baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 48
Pharmacokinetics (PK): Area Under the Curve (AUC) of LY3841136 | Baseline, Week 48
PK: Maximum Concentration (Cmax) of LY3841136 | Baseline, Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (52):
- United States (48):
  - The Institute for Liver Health II dba Arizona Clinical Trials - Mesa, Chandler, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - The Institute for Liver Health II dba Arizona Liver Health-Tucson, Tucson, Arizona
  - NorCal Medical Research, Inc, Greenbrae, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Medical Research Partners, Ammon, Idaho
  - Great Lakes Clinical Trials - Andersonville, Chicago, Illinois
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - NorthShore University Health System, Skokie, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - Knownwell, Needham, Massachusetts
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Headlands Research - Detroit, Southfield, Michigan
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Headlands Llc, Springfield, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Dent Neurologic Institute, Amherst, New York
  - Velocity Clinical Research, Syracuse, East Syracuse, New York
  - North Suffolk Neurology, Port Jefferson Station, New York
  - Rochester Clinical Research, LLC, Rochester, New York
  - Medication Management, Greensboro, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Lucas Research, Inc, Morehead City, North Carolina
  - Lucas Research, Inc., New Bern, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Quality Medical Research, Nashville, Tennessee
  - IMA Clinical Research Austin, Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Tekton Research - Fredericksburg Road, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Texas Valley Clinical Research, Weslaco, Texas
  - Spectrum Medical, Inc., Danville, Virginia
  - Central Washington Health Services Association d/b/a Confluence Health, Wenatchee, Washington
- Argentina (4):
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study to Investigate Weight Management With LY3841136 and Tirzepatide (LY3298176), Alone or in Combination, in Adult Participants With Obesity or Overweight With Type 2 Diabetes — https://trials.lilly.com/en-US/trial/533180